CLINICAL TRIAL: NCT06284811
Title: Effects of Massage and Percussion Therapy on Muscle Viscoelastic Properties, DOMS and Vertical Jump Performance Parameters
Brief Title: Massage and Percussion Therapy on Muscle and Performance Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Collaborators: Istanbul Aydın University (Other); Biruni University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 050.06.04/155
Record Dates: First submitted 2024-01-24; First posted 2024-02-29 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2024-02

CONDITIONS: Healthy
Keywords: percussion therapy; physically active; Massage; viscoelastic properties; DOMS; vertical jump performance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Percussion therapy group (Experimental): After exercises completed, individuals receive percussion therapy on quadriceps for 10 minutes for both sides. Afterwards individuals will be evaluated again.
  Interventions: Behavioral: HIIT Exercise program focusing on quadriceps
- Massage therapy group (Active Comparator): After exercises completed, individuals receive massage therapy on quadriceps for 10 minutes for both sides. Afterwards individuals will be evaluated again.
  Interventions: Behavioral: HIIT Exercise program focusing on quadriceps

INTERVENTIONS:
Behavioral: HIIT Exercise program focusing on quadriceps — Participants will be asked to perform the exercise program that focusing on quadriceps muscle.the participants started to 20-minute HIIT for the lower extremity. The HIIT protocol included static lunch, squats, squat walk, sumo squat, lateral squat walk, front and back lunge, kneel to squat, squat pulses and side lunge exercises. Exercises were performed as 40 seconds exercise and 10 seconds rest. During training, heart rate (HR) was monitored using an activity monitor. All participants completed HIIT Training, after received either percussion therapy or massage therapy according to their randomizations.

SUMMARY:
DOMS, muscle viscoelastic properties, quadriceps strength and vertical jump performance will be evaluated in physically active individuals before the exercise and after the exercise and intervention which is either Swedish massage or Percussion therapy

DETAILED DESCRIPTION:
Intense physical activity affects the biochemical balance of muscle cells by stimulating the accumulation of inorganic phosphate, protons, lactate and free Mg2+. The altered biochemical balance leads to fatigue, resulting in impaired exercise capacity and manifested by a decrease in the intensity and efficiency of muscle work. The optimal balance between training and post-training recovery is one of the main elements to consider due to its impact on muscle strength, physical performance and delayed onset muscle soreness (DOMS).

One such recovery tool which has recently grown in popularity is handheld percussive massage devices (i.e., massage guns). The first commercial massage gun was invented in 2008 and in recent years, there has been an increase in popularity of handheld devices for personal and professional therapeutic use, as well as by physiotherapists, strength and conditioning coaches and athletes to elicit potential performance gains.

Massage is defined as "the mechanical manipulation of body tissues with rhythmic pressure and stroking to promote health and well-being" and is used for recovery, pre-exercise preparation and injury prevention and rehabilitation.

Massage is known to reduce muscle tension; reduce muscle pain, edema and spasm; improve flexibility and range of motion; increase blood flow in the muscle and clear substances such as blood lactate or creatine kinase, and therefore have effects on fatigue.

Rapid recovery of performance is important for both amateur and professional athletes, and scientific studies are needed to prove that massage is an effective tool to improve post-exercise recovery or to promote a faster recovery.

To the best of our knowledge, literature lacks studies that compare percussion therapy and massage therapy effects on recovery, muscle strength and performance post-exercise. The aim of this study will be to examine the effect between percussion massage with a mechanical percussion device and classical Swedish massage after acute exercise.

ELIGIBILITY:
Inclusion Criteria:

* Participants willing to provide informed consent to participate in the study.
* Healthy adults aged between 18 and 30 years.
* No history of musculoskeletal injuries within the past six months.
* No known cardiovascular or respiratory conditions that may affect exercise performance.
* Participants with no previous experience with either massage or percussion therapy.
* International Physical Activity Questionnaire - Short Form questionnaire score above 3000

Exclusion Criteria:

* Any medical condition or history of medical conditions that could affect muscle function or recovery (e.g., chronic pain conditions, autoimmune disorders).
* Individuals taking medications that could influence muscle performance or recovery.
* Any current injuries or pain that may interfere with the ability to perform exercises or receive interventions.
* Known allergies to massage oils or lotions or individuals with skin conditions that may be exacerbated by massage or percussion therapy.
* Participants unwilling or unable to comply with the study protocol.
* Inability to understand the study requirements.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-12-31 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-09-20 (Actual)

PRIMARY OUTCOMES:
Muscle tone/tension(Hz) | 10 weeks
  3 parts of quadriceps(Rektus femoris, Vastus medialis, Vastus lateralis) will be evaluated will be evaluated with Myoton PRO device through holding it on the muscle.
Muscle dynamic stiffness (N/m) | 10 weeks
  3 parts of quadriceps(Rektus femoris, Vastus medialis, Vastus lateralis) will be evaluated will be evaluated with Myoton PRO device through holding it on the muscle.
Muscle elasticity (log) | 10 weeks
  3 parts of quadriceps(Rektus femoris, Vastus medialis, Vastus lateralis) will be evaluated will be evaluated with Myoton PRO device through holding it on the muscle.
DOMS | 10 weeks
  DOMS will be evaluated with Visual Analogue Score, minimum value of 0, maximum value of 10. Visual Analogue Score, highest(10) will be for the soreness at its highest, and lowest(0) for no soreness at all.
Vertical Jump Performance | 10 weeks
  Individual's vertical jump performance will be evaluated in cm.
Quadriceps isometric strength | 10 weeks
  Quadriceps isometric strength will be evaluated with hand held dynamometer

CONTACTS AND LOCATIONS:
Locations (1):
- Acibadem University, Istanbul, Ataşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garcia-Sillero M, Benitez-Porres J, Garcia-Romero J, Bonilla DA, Petro JL, Vargas-Molina S. Comparison of Interventional Strategies to Improve Recovery after Eccentric Exercise-Induced Muscle Fatigue. Int J Environ Res Public Health. 2021 Jan 14;18(2):647. doi: 10.3390/ijerph18020647. PMID 33466606
- [Background] Sams L, Langdown BL, Simons J, Vseteckova J. The Effect Of Percussive Therapy On Musculoskeletal Performance And Experiences Of Pain: A Systematic Literature Review. Int J Sports Phys Ther. 2023 Apr 1;18(2):309-327. doi: 10.26603/001c.73795. eCollection 2023. PMID 37020441
- [Background] Chwala W, Pogwizd P, Rydzik L, Ambrozy T. Effect of Vibration Massage and Passive Rest on Recovery of Muscle Strength after Short-Term Exercise. Int J Environ Res Public Health. 2021 Nov 7;18(21):11680. doi: 10.3390/ijerph182111680. PMID 34770194
- [Background] Akinci B, Zenginler Yazgan Y, Altinoluk T. The effectiveness of three different recovery methods on blood lactate, acute muscle performance, and delayed-onset muscle soreness: a randomized comparative study. J Sports Med Phys Fitness. 2020 Mar;60(3):345-354. doi: 10.23736/S0022-4707.19.10142-9. Epub 2019 Oct 28. PMID 31684705
- [Background] Canbulut A, Kıyak G, Ercan S, Çetin C. Acute effect of percussion massage applied on quadriceps with Hypervolt device on range of motion and performance. Spor Hekimliği Dergisi. 2023;58(2):055-60.
- [Background] Menek MY, Menek B. Effects of percussion massage therapy, dynamic stretching, and static stretching on physical performance and balance. J Back Musculoskelet Rehabil. 2024;37(1):183-193. doi: 10.3233/BMR-230069. PMID 37661870
- [Background] Leabeater AJ, Clarke AC, James L, Huynh M, Driller M. Under the Gun: Percussive Massage Therapy and Physical and Perceptual Recovery in Active Adults. J Athl Train. 2024 Mar 1;59(3):310-316. doi: 10.4085/1062-6050-0041.23. PMID 37248364